CLINICAL TRIAL: NCT00556699
Title: An Open-Label, Phase Ib Study of the Safety, Pharmacokinetics, and Activity of the Anti-CD40 Monoclonal Antibody SGN-40 Administered in Combination With Rituximab in Patients With CD20-Positive, Follicular and Marginal Zone B-Cell Non-Hodgkin's Lymphoma Who Have Relapsed Following Previous Rituximab Therapy
Brief Title: A Study of SGN-40 in Combination With Rituximab in Patients With CD20-Positive, Follicular and Marginal Zone B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACF4325g
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2011-11

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NHL; Rituxan; anti-CD40
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; dacetuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab; Drug: SGN-40

INTERVENTIONS:
Drug: rituximab — Escalating intravenous repeating dose
Drug: SGN-40 — Escalating intravenous repeating dose

SUMMARY:
This is an open-label, multicenter Phase Ib study designed to evaluate the safety, pharmacokinetics, and preliminary efficacy of SGN-40 when combined with rituximab in patients with relapsed CD20-positive, follicular or marginal zone NHL who have received at least one prior rituximab-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of histologically confirmed CD20-positive, follicular NHL or marginal zone NHL
* At least one previous treatment with rituxan monotherapy or a rituximab-containing regimen
* Measurable disease
* Either fresh or archived tumor specimen must be available for central confirmation of diagnosis and correlative studies
* Life expectancy of > 3 months
* For patients of reproductive potential, use of a reliable means of contraception

Exclusion Criteria:

* Chemotherapy or radiotherapy within 28 days of Day 1
* Prior treatment with a monoclonal antibody directed against CD40
* Radioimmunotherapy or immunotherapy with a monoclonal antibody other than rituximab within 3 months of Day 1
* Prior treatment with an investigational drug within 28 days of Day 1
* Prior allogeneic bone marrow transplant
* Prior autologous hematopoietic stem cell transplant within 12 weeks of Day 1
* Concurrent systemic corticosteroid therapy
* Prior anaphylactoid or other serious reaction to rituximab that resulted in hospitalization or discontinuation of therapy, or both
* Evidence of clinically detectable ascites on Day 1
* Other invasive malignancies within 3 years prior to Day 1 except for adequately treated basal cell or squamous cell skin cancer, in situ carcinoma of the cervix, in situ breast cancer, in situ prostate cancer, or other cancer of which the patient has been disease-free for at least 3 years
* History or evidence on physical examination of CNS disease
* Active infection requiring parenteral antibiotics within 14 days of Day 1
* Major surgical procedure (excluding lymph node biopsy) or significant traumatic injury within 28 days prior to Day 1
* Pregnancy (positive pregnancy test) or lactation
* Serious, nonhealing wound, ulcer, or bone fracture
* Clinically significant cardiovascular disease, congestive heart failure, serious cardiac arrhythmia requiring medication within 1 year prior to Day 1. Grade II or greater peripheral vascular disease at study entry.
* Known human immunodeficiency virus (HIV) infection
* Known serious medical conditions, including cirrhosis, hepatitis C infection, and chronic obstructive or chronic restrictive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities in order to determine the maximum tolerated dose | Length of study

SECONDARY OUTCOMES:
Changes in vital signs, physical examination findings, and clinical laboratory results | Length of study
Incidence, nature, and severity of adverse events | Length of study
Pharmacokinetic parameters | Length of study
Patient's best response as assessed by the investigator | Length of study
Duration of response | Length of study
Event-free survival | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Hurst, M.D., Study Director — Genentech, Inc.